CLINICAL TRIAL: NCT07061470
Title: RestEaze: A Novel Wearable Device and Mobile Application to Improve the Diagnosis and Management of Restless Sleep in Pediatric Patients With Attention Deficit/Hyperactivity Disorder, Phase II
Brief Title: A Clinical Trial of Iron Supplementation for Youth With ADHD and Restless Sleep
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00511528
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: ADHD; Sleep Problems
Keywords: ADHD; iron supplements; sleep; restlessness; attention; restless legs syndrome
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias; Psychomotor Agitation; Restless Legs Syndrome | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron supplementation arm (Experimental): Participants in the iron supplementation arm will receive 3 months of iron supplementation treatment
  Interventions: Dietary Supplement: Ferrous Sulfate
- Placebo arm (Placebo Comparator): Participants in the placebo arm will receive 3 months of placebo treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — Dosing of the iron supplement will be based on weight.
  Arms: Iron supplementation arm
Other: Placebo — Placebo pills will be provided to participants in the placebo arm
  Arms: Placebo arm

SUMMARY:
The goal of this clinical trial is to learn if iron supplementation works to restless sleep in youth with ADHD. A second goal is to learn if iron supplementation helps to ease ADHD symptoms. The main questions that this trial aims to answer are:

Does 3 months of iron supplementation treatment improve parent- and youth self-reported sleep difficulties more than placebo? Does 3 months of iron supplementation treatment improve sleep as measured by actigraphy more than placebo? Does 3 months of iron supplementation treatment improve parent-reported and/or objectively measured attention more than placebo?

Researchers will compare over-the-counter iron supplementation treatment to a placebo (a look-alike substance that contains no drug) to see if iron supplementation works to treat sleep difficulties in youth with ADHD.

Participants will:

* Take iron supplements every day for 3 months
* Visit the clinic once before treatment begins and once at the end of treatment to complete tests and rating scales related to sleep and attention
* Wear motion-monitoring leg bands while sleeping for one 2-week period before treatment begins and one 2-week period at the end of treatment

DETAILED DESCRIPTION:
Study Population Seventy youth (n=70) will be recruited for participation in the proposed study. Youth meeting eligibility criteria will be recruited through Kennedy Krieger Institute's Sleep Disorders Clinic and Center for Neuropsychological and Psychological Assessment (CNaP). Recruitment will be accomplished by posting flyers with study information at the clinics, by reviewing medical record information of upcoming patients to determine potential eligibility, and by asking clinicians to discuss the study with their patients who may be eligible and their caregivers.

Study Design A double-blind, placebo-controlled randomized superiority trial design will be used in this study. Seventy participants will be assigned to treatment and control conditions using permuted block randomization, based on sequential enrollment and equal allocation to study conditions. Both the participant and members of the study team involved in data collection or outcomes assessment will be blinded to the participant's treatment assignment. The treatment interval for the study will be 3 months, which has been sufficient in previous studies to allow for treatment effects to be observed. Pre-treatment and post-treatment, the following data will be collected for each participant:

1) a complete iron blood panel; 2) 14 consecutive nights of actigraphy monitoring using the RestEaze device at home; 3) parent- or self-ratings of sleep quality over the same 14 nights on which the device is worn; 4) ratings of ADHD symptoms(ADHD-RS-V5) completed by parent and teacher; 5) ratings of sleep problems completed by parent; and 6) neuropsychological testing of attention.

Study Treatment Iron supplementation. The NatureMade brand of iron supplement will be administered to all participants in the treatment condition to minimize variability in concentration of the active ingredients across brands/preparations of iron supplements. This brand of iron supplement is independently verified by United States Pharmacopeia (USP), which conducts rigorous evaluation and monitoring of dietary supplements to ensure that they contain the necessary ingredients at the dosages that are claimed by the manufacturer. Dosing will be determined for each participant by the study physician based on weight. All NatureMade pills will be over encapsulated by the Johns Hopkins Investigational Drug Service to ensure treatment blinding for patients. At the conclusion of study participation, participants will work with their physician to determine whether iron supplementation should be continued.

Placebo. Placebo pills will be manufactured by the Johns Hopkins Investigational Drug Service to match the appearance of the over encapsulated NatureMade pills. At the conclusion of the study, participants assigned to the placebo condition whose blood ferritin levels remain under 50ng/mL will be offered a free 3-month supply of the NatureMade active iron treatment.

Treatment adherence. To monitor treatment adherence, all pills (iron and placebo) will be provided to participants in MEMS cap smart pill bottles. Each plain bottle will be labeled with the participant's name and directions for use and will have a MEMS cap which records the date and time each time the cap is removed from the bottle. These data will be stored, linked to the participant's ID number, in the smart pill bottle software and then downloaded to a secure local server within Kennedy Krieger Institute. These data will allow for daily monitoring of treatment adherence by study personnel, which will provide the opportunity for study personnel to reach out to the participant to encourage compliance or troubleshoot any problems throughout each child's study participation. Participants will be removed from the study prior to completion if they experience significant adverse effects of the treatment, if they do not adhere to treatment or initiate other confounding treatments, or at the request of the patient/family.

Measurement of Peripheral Iron Concentrations. Peripheral iron concentrations will be obtained as part of routine clinical care pre- and post-iron supplementation. Standard indicators of iron availability and storage will be tested with a fasting complete blood count (CBC), serum iron, serum ferritin, total iron binding capacity (TIBC) and transferrin level.

Study Outcomes Study outcomes are reported in the Outcome Measures section.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed with ADHD
* have blood ferritin level below 50ng/mL
* have parent- or self-reported restless sleep

Exclusion Criteria:

* presence of any chronic medical or genetic condition that could impact iron metabolism
* presence of moderate to severe Obstructive Sleep Apnea
* having received Iron supplementation treatment within the past 3 months
* having blood ferritin level indicative of anemia that requires immediate treatment

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | Sleep efficiency will be assessed nightly for 2 weeks before treatment begins and then again for 2 weeks at the end of treatment.
  Sleep efficiency refers to the proportion of time in bed spent sleeping and is measured via actigraphy monitoring. Higher scores indicate more efficient/better sleep.

SECONDARY OUTCOMES:
Total sleep time | These will be assessed nightly for a period of 2 weeks before treatment begins and then again for 2 weeks at the end of treatment.
  Total sleep time in minutes as measured by actigraphy. Higher scores indicate more time asleep.
Wake after sleep onset | These will be assessed nightly for a period of 2 weeks before treatment begins and then again for 2 weeks at the end of treatment.
  Number of minutes spent awake between falling asleep at night and getting up in the morning, as measured by actigraphy. Higher scores on this measure are indicative of greater difficulty staying asleep through the night.
Latency to sleep onset | Assessed nightly for a period of 2 weeks before treatment begins and then again for 2 weeks at the end of treatment.
  Number of minutes from laying down in bed for the night to falling asleep, measured by actigraphy. Higher scores on this measure will indicate longer times to fall asleep.
Attention Deficit Hyperactivity Disorder-Rating Scale-V, parent version | Completed at baseline and again within 2 weeks post-treatment.
  Parent rating of child's ADHD symptoms; raw scores will be calculated by summing all items and will range from 0-54; higher scores indicate more severe ADHD symptoms.
Attention Deficit Hyperactivity Disorder-Rating Scale-V, self report | Completed at baseline and again within 2 weeks post-treatment.
  Youth self-report of ADHD symptoms; raw scores will be calculated by summing all items and will range from 0-54; higher scores indicate more severe ADHD symptoms.
Conners Continuous Performance Test (CPT), 3rd edition | Completed at baseline and again within 2 weeks post-treatment.
  This computer-administered go/no-go test was designed to measure response preparation, sustained attention, and inhibitory control. Ex-Gaussian decomposition of response time variability will the primary indicator of sustained attention, and number of omission and commission errors will serve as indices of cognitive control. The CPT-3 is normed for children ages 8 and up and takes 14 minutes to complete. T-scores (min = 10, max = 90) comparing the participant's performance to normative data will be used. Higher T-scores indicate worse sustained attention, response preparation, and inhibitory control.
Children's Sleep Habits Questionnaire | Completed at baseline and again within 2 weeks post-treatment.
  The CSHQ is a 45-item parent-report questionnaire assessing eight domains of a child's sleep: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep-Disordered Breathing, and Daytime Sleepiness. The measure has demonstrated adequate psychometric properties; except for criterion-related validity. These common areas of concern for children's sleep will be rated by parents on a 3-point Likert scale once pre-treatment and again post-treatment. Ratings on this measure will be used to evaluate sleep-related concerns other than restlessness, as well as change in these concerns with treatment. The total raw score will be calculated by summing all item scores (minimum = 0, maximum = 135) with higher scores indicating more sleep problems.
Sleep Quality Scale | Completed daily for 2 weeks at baseline and then again daily for 2 weeks post-treatment.
  The SQS is a single item measure of overall sleep quality. Respondents are asked to answer to the question "How would you rate your sleep quality overall last night?" using a 0-10 scale where 0 represents "terrible," 1-3 represent "poor," 4-6 represent "fair," 7-9 represent "good," and 10 represents "excellent." Participants in the present study will be asked to rate their sleep each night during the 14 nights on which they are wearing the RestEaze bands pre- and post- treatment.
Wechsler Intelligence Measures, Cancellation Subtest | Completed at baseline and again within 2 weeks post-treatment.
  The Cancellation subtest from the Wechsler Intelligence measures will be used as an index of focused attention. This subtest requires the child to mark target objects and ignore distracters in both a structured and a random array. It takes approximately 5 minutes to administer. Age-appropriate versions of the same task are available for children ages 6-16 (WISC-V), and ages 17+ (WAIS-IV). Norm-referenced scaled scores will be reported (min = 1, max = 19), with higher scores indicating better focused attention.
NIH Toolbox Flanker Task | Completed at baseline and again within 2 weeks post-treatment.
  The flanker task is a measure of attention and inhibitory control. For this task, the child is required to focus attention on a specified stimulus, while inhibiting attention to stimuli positioned on either side of the specified stimulus. The age-adjusted scaled score for this task combines reaction time and accuracy. This task takes less than 10 minutes to administer and is appropriate for children ages 3 and up. Norm-referenced Standard Scores (min = 55, max = 145) will be reported, with higher scores indicating better cognitive flexibility.
NIH Toolbox Dimensional Change Card Sort task | Completed at baseline and again within 2 weeks post-treatment.
  This task is a measure of cognitive flexibility and control. It requires the child to matcha series of pictures first on one dimension (e.g., color), then on another dimension (e.g., shape) with only accuracy feedback as a guide after each trial (no explicit statement of the matching rule). The age-adjusted scaled score for this task combines reaction time and accuracy. This task, recommended for children ages 3 and up, takes less than 10 minutes to administer. Norm-referenced Standard Scores (min = 55, max = 145) will be reported, with higher scores indicating better cognitive flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Pritchard, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No